CLINICAL TRIAL: NCT05494359
Title: The Diagnostic Value of Various Mass Nitrogen Components Excreting for Oral Gas in Esophagus Cancer
Brief Title: The Diagnostic Value of Nitrogen Element (N) in Esophagus Cancer
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, Professor of Surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: Nitrogen element
Record Dates: First submitted 2022-08-07; First posted 2022-08-10 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; Nitrogen mass-charge ratio abundances (NMARs); Diagnosis
MeSH Terms: conditions — Esophageal Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ESCA group: 40 patients of ESCA were included through the diagnosis of gastroscopic biopsy positive.
  Age, gender, esophageal cancer staging, tumor biomarkers and other laboratory test indicators, CT and other imaging examinations results, gastroscope and pathological examinations results have been collected.
  Interventions: Diagnostic Test: The nitrogen isotope
- Health control: 40 healthy people who experienced negative gastroscopy and tumor biomarkers were included as healthy control.
  Age, gender, gastroscope, tumor biomarkers and other laboratory test results have been collected.
  Interventions: Diagnostic Test: The nitrogen isotope
- Reflux esophagitis: 40 patients of reflux esophagitis were included. Age, gender, tumor markers and other laboratory test indicators, gastroscope and pathological examinations results have been collected.
  Interventions: Diagnostic Test: The nitrogen isotope

INTERVENTIONS:
Diagnostic Test: The nitrogen isotope — The nitrogen mass-charge ratio abundances (NMAs) and NMA ratios (NMARs) The nitrogen components of various m/z values in oral gas were detected.

SUMMARY:
The purpose of this study is to determine the diagnostic value of various nitrogen components in oral gas for esophagus cancer (ESCA) .

DETAILED DESCRIPTION:
Less effective diagnostic markers for ESCA can be used in present. Nitrogen elements include a variety of nitrogen components (each corresponding to a specific mass-charge ratio [m/z] value). Stable nitrogen isotope ratios 15 Nitrogen/14 Nitrogen (15 N/14 N) are of particular advantage to understand the metabolic state of cancer cells, since most biochemical reactions involve transfer of nitrogen. Cancerous cells can recycle metabolic ammonium for their growth . The recycling of this ammonium with a low nitrogen isotope ratio (15 N/14 N) may cause cancer tissue to have lower 15 N/14 N than surrounding healthy tissue, and it could diagnose malignancy as well as an avenue for investigation of cancer metabolism.

However, the relationship and diagnostic value between nitrogen excretion from oral gas and ESCA remains unclear. The purpose of this study is to analyze the diagnostic value of various mass nitrogen components excreting for oral gas for ESCA.

ELIGIBILITY:
Inclusion Criteria:

* Esophageal cancer patients (Case): Subject diagnosed with ESCA based on typical clinical symptoms, endoscopic observation of esophageal lesions, and histopathological examination of biopsy specimens obtained from the lesion sites.
* Reflux esophagitis patients (Case control): Subject diagnosed diagnosed with reflux esophagitis based on typical clinical symptoms (e.g., heartburn and acid regurgitation) and endoscopic evidence of esophageal mucosal injury classified according to the Los Angeles classification system (Grade A: mucosal breaks ≤5 mm in length; Grade B: mucosal breaks >5 mm in length but not confluent; Grade C: confluent mucosal breaks involving <75% of the esophageal circumference; Grade D: confluent mucosal breaks involving ≥75% of the esophageal circumference).
* Health people: (Healthy control): no history of malignant tumors within the past five years, normal findings on gastroscopy, with no evidence of esophageal or gastric lesions, no history of gastrointestinal diseases such as gastroesophageal reflux disease (GERD) or Barrett's esophagus, blood counts, tumor biomarkers, and liver and kidney function tests within normal ranges.

Exclusion Criteria:

* Esophageal or gastric surgery
* History of previous upper abdominal surgery
* History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
* History of other malignant disease within past five years
* History of previous neoadjuvant chemotherapy or radiotherapy
* History of unstable angina or myocardial infarction within past six months
* History of cerebrovascular accident within past six months
* Requirement of simultaneous surgery for other disease
* Emergency surgery due to complication (bleeding, obstruction or perforation) caused by cancer
* Pregnant women or breastfeeding
* Unwillingness or inability to consent for the study
* Severe mental disorder
* Unstable vital signs Coagulation dysfunction (INR>1.5)
* Low peripheral blood platelet or using anti coagulation drugs
* Long-term Chinese medicine treatment of unknown drug nature

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 esophageal cancer patients; 40 reflux esophagitis patients; 40 health volunteers
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-11-16 (Actual); Study Completion 2024-11-16 (Actual)

PRIMARY OUTCOMES:
15 Nitrogen/14 Nitrogen (15 N/14 N),28 N/14 N, 29 N/14 N,30 N/14 N, 28 N/ 15 N , 29 N/15 N,30 N/15 N, 28 N/ 16 N , 29 N/16 N, 30 N/16 N,29 N/28 N,30 N/18 N,30 N/29 N ratio. | 1 week
  The normal "Nitrogen" ratio reference interval were 0.18-0.20, 69-78, 122-143, 0.9-1.1, 340-410, 602-747, 4.4-5.6, 390-500 , 700-960, 5.1-7.3, 1.7-1.9, 0.009-0.011, 0.007-0.08, respectively.
The number of 15 Nitrogen, 14 Nitrogen, 16 Nitrogen, 28 Nitrogen, 29 Nitrogen, 30 Nitrogen. | 1 week
  The normal 15 Nitrogen, 14 Nitrogen, 28 Nitrogen, 29 Nitrogen, 30 Nitrogen reference interval were 98000-140000, 98000-140000, 33000-60000, 4090000-4630000, 7100000-8200000, 520000-610000, respectively.
The area under curve value of exhaled mass nitrogen components for esophageal cancer. | 1 week
  Area under curve is the area under the Receiver Operating Characteristic (ROC) curve, serving as a crucial metric for evaluating the performance of classification exhaled nitrogen indicators (nitrogen mass-charge ratio abundances, and nitrogen mass-charge ratio abundances ratios) .
The sensitivity and specificity of exhaled mass nitrogen components for esophageal cancer. | 1 week
  The sensitivity and specificity will be determined by comparing the result to the clinical gold standard gastroscope. They reflect the reliability of the test results.

SECONDARY OUTCOMES:
The differentiation type of the tumor. | 1 week
  The type of differentiation, low, moderate or high by histology
The stage of the cancer. | 1 week
  According to the primary tumor, regional nodes, metastasis classification
The accuracy of exhaled mass nitrogen components for the diagnosis of esophageal cancer stages and invasion. | 1 week
  The ROC curve, sensitivity and specificity of various representative exhaled nitrogen indicators (nitrogen mass-charge ratio abundances, and nitrogen mass-charge ratio abundances ratios) for detecting early-stage (I and II ) and invasion (T1/T2).
The negative and positive predictive value of exhaled nitrogen indicators (nitrogen mass-charge ratio abundances, and nitrogen mass-charge ratio abundances ratios) for detecting ESCA and different subgroups ESCA. | 1 week
  The positive and negative predictive value will be determined based on true positive and false positive, and true negative and false negative, respectively. They reflect the reliability of the test results.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu
  - Wuwei Tumor Hospital, Wuwei, Gansu
  - Clinical Research Centre, The Seventh Affiliated Hospital, Shenzhen, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided
Individuals may be reluctant to divulge health information

REFERENCES:
- [Result] Krishnamurthy RV, Suryawanshi YR, Essani K. Nitrogen isotopes provide clues to amino acid metabolism in human colorectal cancer cells. Sci Rep. 2017 May 31;7(1):2562. doi: 10.1038/s41598-017-02793-y. PMID 28566705
- [Result] Straub M, Sigman DM, Auderset A, Ollivier J, Petit B, Hinnenberg B, Rubach F, Oleynik S, Vozenin MC, Martinez-Garcia A. Distinct nitrogen isotopic compositions of healthy and cancerous tissue in mice brain and head&neck micro-biopsies. BMC Cancer. 2021 Jul 13;21(1):805. doi: 10.1186/s12885-021-08489-x. PMID 34256713